CLINICAL TRIAL: NCT05571072
Title: Opioid Use After Urogynecologic Procedures: Using a Predictive Calculator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Sheyn (Other)
Responsible Party: Sponsor-Investigator, David Sheyn, Associate Professor of Urology, University Hospitals Cleveland Medical Center
Organization: University Hospitals Cleveland Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY20221287
Record Dates: First submitted 2022-10-04; First posted 2022-10-07 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Post Operative Pain; Opioid Use; Prolapse Genital
Keywords: post operative pain; opioid use; urogynecologic surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Opioid Prescription (Active Comparator): Patients will be given a prescription for opioid pain medication to use for acute postoperative pain as would be typical for the attending surgeon performing the surgery.
  Interventions: Other: Standard opioid prescription
- Opioid Calculator Prescription (Experimental): Patients will be a given a prescription for opioid pain medication based on the opioid calculator.
  Interventions: Other: Opioid calculator

INTERVENTIONS:
Other: Opioid calculator — Our research group previously created an Opioid calculator that can be used to predict the number of opioids needed post-operatively based on patient health history and characteristics.
  Arms: Opioid Calculator Prescription
Other: Standard opioid prescription — Patients will receive prescription for post-operative opioids based on what the attending surgeon usually provides.
  Arms: Standard Opioid Prescription

SUMMARY:
The purpose of this study is to determine if the investigators can precisely predict how much pain medication the subjects will need after surgery using a special calculator that was developed for this purpose.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-89
* Able to provide informed consent
* Patients undergoing any of below urogynecologic procedures

Included urogynecologic procedures:

1. Sacrocolpopexy - robotic or laparoscopic

   1. With or without hysterectomy
   2. With or without salpingo-oophorectomy
   3. With or without anterior colporrhaphy
   4. With or without posterior colporrhaphy/perineorrhaphy
   5. With or without midurethral sling
2. Sacrospinous ligament fixation

   1. With or without hysterectomy
   2. With or without salpingo-oophorectomy
   3. With or without anterior colporrhaphy
   4. With or without posterior colporrhaphy/perineorrhaphy
   5. With or without midurethral sling
3. Uterosacral ligament suspension - robotic, laparoscopic, or vaginal

   1. With or without hysterectomy
   2. With or without salpingo-oophorectomy
   3. With or without anterior colporrhaphy
   4. With or without posterior colporrhaphy/perineorrhaphy
   5. With or without midurethral sling
4. Colpocleisis

   1. Lefort colpocleisis
   2. Complete colpectomy with colpocleisis
5. Isolated anterior and/or posterior colporrhaphy

Exclusion Criteria:

* Non-English speakers
* pre-operative diagnosis of cancer
* scheduled for any concurrent non-urogynecologic procedure (ex: abdominoplasty)
* <18 years or >89 years of age
* unable to provide informed consent

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2024-02-17 (Actual); Study Completion 2024-02-17 (Actual)

PRIMARY OUTCOMES:
Change in pain scores measured by team-created pain questionnaires | baseline, 1 week post-op, 2 weeks post-op
  Pain questionnaire is a 2 question survey that ask patients to rate pain on scale of 0 (no pain) to 10 (worst pain) immediately post-op and current. Baseline will be calculated by asking patient's expected post-op pain score.

SECONDARY OUTCOMES:
Change in satisfaction scores measured by team-created questionnaire | 1 week post-op, 2 weeks post-op
  Questionnaire is a 1 question survey that ask patients to rate their satisfaction with their pain control on scale of 0 (totally unsatisfied) to 10 (totally satisfied) immediately post-op and current.
Change in number of opioid tablets remaining measured by team-created questionnaire | 1 week post-op, 2 weeks post-op
  Patients will be asked the number of tablets remaining from their opioid prescriptions.

CONTACTS AND LOCATIONS:
Overall Officials: David Sheyn, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bauer HH, Schlussel MA, Hoffberg EA, Palm KM, Rhodes SP, Wherley SD, Le Neveu M, Sears SB, Rustia GM, Hijaz AK, Mahajan ST, Sammarco AG, Sheyn D. Personalized Prediction of Opioid Demand After Surgery for Pelvic Organ Prolapse: A Randomized Controlled Trial. Obstet Gynecol. 2025 Jun 26;146(2):285-292. doi: 10.1097/AOG.0000000000005969. PMID 40570353